CLINICAL TRIAL: NCT04259424
Title: Priming Upper Extremity Motor Practice With Aerobic Exercise: A Feasibility and Pilot Study
Brief Title: Exercise-primed Upper Extremity Motor Practice in Chronic Stroke
Acronym: PUMP-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Ryan Ross, Post-Doctoral Scholar, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro#00092739
Record Dates: First submitted 2020-01-27; First posted 2020-02-06 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Stroke
Keywords: Rehabilitation; Upper Extremity; Aerobic Exercise; Motor Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: All subjects enrolled will receive the same treatment. Upper extremity motor function outcome measures will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Aerobic Exercise + Upper Extremity Rehabilitation (Experimental): Subjects will receive a total of 18 intervention sessions. In each intervention session, subjects will perform 15 minutes of aerobic exercise on a stationary cycle followed by 200 repetitions of an upper extremity rehabilitation program.
  Interventions: Device: Aerobic Exercise + Duck Duck Punch

INTERVENTIONS:
Device: Aerobic Exercise + Duck Duck Punch — Subjects will perform 15 minutes of aerobic exercise on a recumbent stationary cycle. On each session the target intensity of aerobic exercise will be 70% heart rate reserve.
  Following a 10-minute rest break subjects will perform 200 repetitions on an upper extremity rehabilitation game called Duck Duck Punch (DDP). Duck Duck Punch is an interactive game with an old school carnival theme. DDP is unique as it uses Microsoft Kinect skeletal tracking technology to assess movement performance. The participant sits in front of the Microsoft Kinect and controls a virtual arm with his/her physical arm; reaching forward to "punch" virtual ducks. A therapist will oversee the subject's safety and progress during DDP. DDP will be dosed based on the number of repetitions performed. A repetition is recorded when the player moves his/her arm so that the avatar leaves a start position. The goal dose for subjects will be 200 repetitions per DDP session.

SUMMARY:
The purpose of this project is to establish initial feasibility and tolerability of a combined aerobic exercise (AEx) and upper extremity motor practice intervention on upper extremity (UE) function in chronic stroke survivors. This novel intervention pairs AEx with a virtual reality-based upper extremity rehabilitation game, Duck Duck Punch (DDP). AEx has been shown to improve overall brain function and promote a healthy brain environment; thus it may serve as an effective 'primer' and enhance the effects of DDP. Movement-based priming for rehabilitation involves performing movement or exercise before, or simultaneous to, an intervention with the goal of improving the effectiveness of the intervention. AEx combined with UE rehabilitation can improve UE function and self-reported health status in chronic stroke survivors. However, gaps remain regarding the clinical applicability of an AEx priming session and the mechanisms contributing to changes in UE functions in response to AEx-primed UE rehabilitation. Therefore, the aim of this project is to: 1) demonstrate the feasibility of pairing AEx + DDP in stroke survivors; 2) quantify the magnitude of the effect of the AEx + DDP intervention on UE function; 3) examine relationship of biomarkers of the nervous system and response to AEx + DDP.

DETAILED DESCRIPTION:
With a surviving cohort of nearly 7 million individuals, stroke is the leading cause of long-term disability in the United States. Of the ~795,000 new strokes occurring annually, approximately 2/3rds of survivors will have some degree of long term disability. The prevalence of post-stroke disability coupled with the fact that more people are surviving stroke reflects an increasing need to develop effective rehabilitation strategies aimed at reducing disability and improving quality of life for the millions of stroke survivors, their families and caregivers.

The overwhelming majority of stroke survivors, >75%, exhibit upper extremity (UE) hemiparesis, and only 15% will recover fully. Furthermore, residual UE impairment is closely linked to long-term disability and reduced quality of life. Current meta-analytic evidence supports virtual reality stroke rehabilitation interventions for improving UE function suggesting that this is a promising area for further therapeutic development.

Duck Duck Punch (DDP) is an interactive computer game deliberately designed to enhance UE movement quality via individualized progressive movement practice along with an array of performance metrics allowing for within-session feedback on movement performance. Although response to UE virtual reality rehabilitation interventions, such as DDP, involves a multitude of factors, neuroplastic changes are a primary mechanism underlying functional recovery. Thus, pairing DDP with a priming intervention to facilitate a 'neuroplastic-friendly' environment may make the CNS more amenable, and enhance response to DDP rehabilitation and ultimately improve outcomes.

Aerobic exercise (AEx) training has positive benefits on overall brain function including enhanced global cognition, executive function, and processing speed and attention in healthy, older adults. Additionally, a single session of AEx acutely improves motor memory and learning in younger, healthy adults. Although AEx has been used to improve cardiovascular function following stroke, its neurofacilitatory effects in stroke have yet to be tested empirically. Candidate mechanisms through which AEx enhances brain function and motor learning include changes in circulating brain-derived neurotrophic factor (BDNF) and corticomotor excitability. BDNF is believed to play an integral role in several neuroplastic processes and promotes the strengthening of synaptic connections, i.e. long-term potentiation (LTP) and current research indicates that AEx can acutely and chronically increase circulating BDNF. Corticomotor excitability (CME) is often used as an indicator of LTP-like neuroplasticity and may underlie improvements in motor memory and learning. Similarly to BDNF, AEx can acutely enhance corticomotor excitability in control and chronic stroke subjects. Facilitating central nervous system function provides rationale to determine the role of AEx in 'prime' the brain for a subsequent intervention to maximize neuroplastic potential.

Movement-based priming for neurorehabilitation involves performing movement or exercise before, or concurrent to, a therapeutic intervention with the goal of improving the efficacy of the therapeutic intervention. Emerging evidence supports AEx as a potential priming tool for UE stroke rehabilitation. AEx combined with UE task training can improve UE function and self-reported health status in chronic stroke survivors. Despite the promising results, there are gaps in the literature involving: 1) the clinical applicability of an AEx priming session; and 2) mechanisms contributing to changes in UE functions in response to AEx-primed UE rehabilitation. Addressing these gaps will be necessary to develop an AEx primer that is potent and time efficient, with respect to current clinical models. Therefore, the purpose of this pilot proposal will be to establish initial feasibility and tolerability benchmarks via the following aims:

1. Demonstrate the feasibility of pairing AEx + DDP in stroke survivors with UE hemiparesis
2. Quantify the magnitude of the effect of the AEx + DDP intervention on UE impairment and function
3. Examine the relationship of biomarkers of neuroplasticity (BDNF and corticomotor excitability) and response to AEx + DDP

To accomplish these aims, chronic stroke survivors with moderate UE hemiparesis will undergo 18 sessions of AEx + DDP training. Each week, for six weeks, subjects will undergo three sessions of AEx + DDP. During each session subjects will complete 15 minutes of aerobic exercise followed by 200 repetitions of DDP. Assessment of UE function and biomarkers of neuroplasticity will be assessed before and after the AEx + DDP intervention.

ELIGIBILITY:
Inclusion Criteria:

* experienced unilateral stroke at least 6 months, but no more than 120 months prior
* voluntary shoulder flexion of the affected arm ≥20° with simultaneous elbow extension ≥10°
* moderate arm movement impairment (UE Fugl-Meyer Assessment > 21 but < 52 points
* passive range of motion in paretic shoulder, elbow, wrist, thumb and fingers within 20 degrees of normal
* 21-90 years of age
* ability to communicate as per the therapists' judgement at baseline testing
* ability to complete and pass an exercise tolerance test

Exclusion Criteria:

* lesion in brainstem/cerebellum as these may interfere with visual-perceptual/cognitive skills needed for motor re-learning
* presence of other neurological disease that may impair motor learning skills
* orthopedic condition or impaired corrected vision that alters reaching ability (e.g., prior rotator cuff tear without full recovery)
* paretic arm pain that interferes with reaching
* unable to understand or follow 3-step directions
* severe cognitive impairment (Montreal Cognitive Assessment score <22)
* severe aphasia
* inability to read English
* history of congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during ADL's
* Severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest
* history of, or current, depression and for brain stimulation procedures only
* women of child-bearing potential
* electronic or metallic implants
* history of seizures

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gregory, PhD, PT, Study Director — Medical University of South Carolina
Locations (1):
- Stroke Recovery Research Center, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerobic Exercise + Upper Extremity Rehabilitation: Subjects will receive a total of 18 intervention sessions. In each intervention session, subjects will perform 15 minutes of aerobic exercise on a stationary cycle followed by 200 repetitions of an upper extremity rehabilitation program.
  Aerobic Exercise + Duck Duck Punch: Subjects will perform 15 minutes of aerobic exercise on a recumbent stationary cycle. On each session the target intensity of aerobic exercise will be 70% heart rate reserve.
  Following a 10-minute rest break subjects will perform 200 repetitions on an upper extremity rehabilitation game called Duck Duck Punch (DDP). Duck Duck Punch is an interactive game with an old school carnival theme. DDP is unique as it uses Microsoft Kinect skeletal tracking technology to assess movement performance. The participant sits in front of the Microsoft Kinect and controls a virtual arm with his/her physical arm; reaching forward to "punch" virtual ducks. A therapist will oversee the subject's safety and progress during DDP. DDP will be dosed based on the number of repetitions performed. A repetition is recorded when the player moves his/her arm so that the avatar leaves a start position. The goal dose for subjects will be 200 repetitions per DDP session.
Period: Overall Study
Arm/Group | Aerobic Exercise + Upper Extremity Rehabilitation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aerobic Exercise + Upper Extremity Rehabilitation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper Extremity Impairment as Assessed by the Fugl-Meyer Assessment - Upper Extremity
Description: The FMA-UE is a 33-item measure of upper extremity impairment; however, the 3 items testing reflex response will not be administered because they do not measure a voluntary movement construct. Each item will be scored on a 3-point rating scale (0=unable, 1=partial 2=near normal performance), item ratings will be summed and reported out of 60 points so that larger numbers indicate greater upper extremity motor ability.
Time Frame: Pre and post intervention, approximately 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise + Upper Extremity Rehabilitation
Number analyzed (Participants) | 10
units on a scale | 2.6 (5.2)
Statistical Analysis 1: Comparison: Aerobic Exercise + Upper Extremity Rehabilitation; Test type: Other; p = .15, t-test, 2 sided

2. Secondary Outcome: Change in Upper Extremity as Assessed by the Wolf Motor Function Test
Description: The WMFT is a 15-item measure of UE functional ability. Performance of each item will be timed (seconds) and the average time to perform items will be reported so that lower values indicate greater UE function.
Time Frame: Pre and post intervention, approximately 6 weeks
Population: Change in Wolf Motor Function Test - Time
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Aerobic Exercise + Upper Extremity Rehabilitation
Number analyzed (Participants) | 10
seconds | .1 (17.6)

3. Secondary Outcome: Change in Physical Function and Health-related Quality of Life as Assessed by Stroke Impact Scale
Description: The SIS-hand consists of 5-items regarding difficulty of paretic hand use during everyday tasks during the previous two weeks. Items will be rated on a 5-point scale (5=not difficult, 1=cannot do) and reported as an average item rating. The SIS-recovery subtest is a single-item in which the participant rates his/her perceived post-stroke recovery from 0%-100% recovered.
Time Frame: Pre and post intervention, approximately 6 weeks
Population: Change in Stroke Impact Scale - Recovery subtest, Change in SIS-hand subtest.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise + Upper Extremity Rehabilitation
Number analyzed (Participants) | 10
units on a scale
  SIS - Recovery | 8.5 (10.6)
  SIS - Hand | -0.5 (6.0)

4. Other Pre Specified Outcome: Change in Neuroplastic Potential as Assessed by Paired Associative Stimulation
Description: Participants' neuroplastic potential will be assessed with a plasticity-inducing paradigm called Paired Associative Stimulation (PAS). Briefly, PAS utilizes a repeated and timed peripheral nerve stimulation combined with transcranial magnetic stimulation (TMS) of the contralateral motor cortex to induce motor cortex plasticity. Prior to- and after PAS, corticomotor excitability (CME) is assessed via motor evoked potentials (MEP) which are obtained by single pulse TMS and electromyography (EMG) of a contralateral peripheral muscle.
Time Frame: Pre and post intervention, approximately 6 weeks
Population: Relative change in Post-PAS MEP amplitude from pre-intervention
Measure: Mean (Standard Deviation); unit: percentage of change in MEP amplitude
Arm/Group | Aerobic Exercise + Upper Extremity Rehabilitation
Number analyzed (Participants) | 7
percentage of change in MEP amplitude | 2.2 (34)

5. Other Pre Specified Outcome: Assessment of Peripheral Brain-derived Neurotrophic Factor
Description: Blood specimens will be obtained immediately before and after AEx on three separate occasions (sessions 1, 9, and 18). Briefly, an intravenous catheter will be placed in a superficial forearm vein at the beginning of the experimental session and will be maintained patent using an isotonic saline solution. Baseline blood samples will be drawn immediately before exercise commences. Immediate post-exercise blood samples will be taken within sixty seconds of exercise completion while the participant remains seated in the cycle ergometer.
Time Frame: Pre and post aerobic exercise on intervention sessions 1, 9, and 18. Each aerobic exercise session will be 15 minutes
Population: Change in peripheral BDNF following aerobic exercise (Post aerobic exercise BDNF - Pre aerobic exercise BDNF)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Aerobic Exercise + Upper Extremity Rehabilitation
Number analyzed (Participants) | 10
ng/ml
  Session 1: number analyzed (Participants) | 8
  Session 1 | -4.7 (8)
  Session 9 | -3.2 (13.5)
  Session 18 | -2.3 (7.2)

ADVERSE EVENTS:
Time Frame: Data was collected for each participant through study completion, an average of approximately 8 weeks.
Arm/Group | Aerobic Exercise + Upper Extremity Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise + Upper Extremity Rehabilitation (N=10)
Dehydration (General disorders) | 1 (1) — Participant was treated in the emergency department for dehydration and released. This was an unanticipated problem as it was unexpected, however the event does not appear to be related to study procedures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT04259424/Prot_SAP_002.pdf
  • Informed Consent Form (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT04259424/ICF_001.pdf